CLINICAL TRIAL: NCT03890367
Title: Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine Versus Nimenrix® or NeisVac-C® in Healthy Toddlers 12 to 23 Months of Age
Brief Title: Study on a Quadrivalent Meningococcal Conjugate Vaccine (MenACYW Conjugate Vaccine) Compared to Two Meningococcal Reference Vaccines in European Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MEQ00065; 2018-003790-10 (EudraCT Number); U1111-1217-2456 (Other: UTN)
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Results first posted 2021-10-06 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Meningococcal Immunisation (Healthy Volunteers)
MeSH Terms: interventions — meningococcal group A polysaccharide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind: the participant (or legally acceptable representative), and the Investigator remained unaware of the treatment assignments throughout the study. An unblinded vaccine administrator administered the appropriate vaccine but was not involved in safety data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: MenACYW Conjugate Vaccine (Experimental): Healthy, toddlers aged 12 to 23 months received a single dose of MenACYW Conjugate vaccine on Day 0.
  Interventions: Biological: Meningococcal polysaccharide (serogroups A, C, Y, and W) tetanus toxoid Conjugate vaccine
- Group 2: Nimenrix® Vaccine (Active Comparator): Healthy, toddlers aged 12 to 23 months received a single dose of Nimenrix® vaccine on Day 0.
  Interventions: Biological: Meningococcal polysaccharide group A, C, W-135 and Y Conjugate vaccine
- Group 3: NeisVac-C® Vaccine (Active Comparator): Healthy, toddlers aged 12 to 23 months received a single dose of NeisVac-C® vaccine on Day 0.
  Interventions: Biological: Meningococcal group C polysaccharide Conjugate vaccine adsorbed

INTERVENTIONS:
Biological: Meningococcal polysaccharide (serogroups A, C, Y, and W) tetanus toxoid Conjugate vaccine — Pharmaceutical form: Liquid solution for injection Route of administration: Intramuscular
  Other Names: MenACYW Conjugate vaccine
  Arms: Group 1: MenACYW Conjugate Vaccine
Biological: Meningococcal polysaccharide group A, C, W-135 and Y Conjugate vaccine — Pharmaceutical form: Powder and solvent for suspension for injection Route of administration: Intramuscular
  Other Names: Nimenrix®
  Arms: Group 2: Nimenrix® Vaccine
Biological: Meningococcal group C polysaccharide Conjugate vaccine adsorbed — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Other Names: NeisVac-C®
  Arms: Group 3: NeisVac-C® Vaccine

SUMMARY:
Primary Objective:

To demonstrate:

* the non-inferiority of the seroprotection rate (antibody titers greater than or equal to [>=] 1:8) to meningococcal serogroup C following the administration of MenACYW Conjugate or Nimenrix® as measured by serum bactericidal assay using human complement (hSBA). If this non-inferiority was demonstrated, then
* the non-inferiority of the antibody response (geometric mean titers [GMT]). If this non-inferiority was demonstrated, then
* the superiority of the antibody response (GMT). If this superiority was demonstrated, then
* the superiority of the seroprotection rate.

Or to demonstrate:

* the non-inferiority of the seroprotection rate (antibody titers >= 1:8) to meningococcal serogroup C following the administration of MenACYW Conjugate or NeisVac-C® as measured by serum bactericidal assay using baby rabbit complement (rSBA). If this non-inferiority was demonstrated, then
* the non-inferiority of the antibody response (GMT). If this non-inferiority was demonstrated, then
* the superiority of the antibody response (GMT).

Secondary Objective:

To demonstrate:

* the non-inferiority of the seroprotection rate (antibody titers >= 1:8) to meningococcal serogroup C following the administration of MenACYW Conjugate vaccine or Nimenrix® as measured by rSBA. If this non-inferiority was demonstrated, then
* the non-inferiority of the antibody response (GMT). If this non-inferiority was demonstrated, then
* the superiority of the antibody response (GMT).

Or to demonstrate:

* the non-inferiority of the seroprotection rate (antibody titers >= 1:8) to meningococcal serogroup C following the administration of MenACYW Conjugate vaccine or NeisVac-C® as measured by hSBA. If this non-inferiority was demonstrated, then
* the non-inferiority of the antibody response (GMT). If this non-inferiority was demonstrated, then
* the superiority of the antibody response (GMT) .

DETAILED DESCRIPTION:
Study duration per participant was approximately 30 days including: 1 day of screening and vaccination, a phone call and a safety-follow up/end of study visit at Day 8 and Day 30 after vaccine administration, respectively.

Safety assessment included solicited reactions within 7 days after vaccination, unsolicited adverse events up to 30 days after vaccination, serious adverse events and adverse event of special interest throughout the study.

ELIGIBILITY:
Inclusion criteria :

* Aged 12 to 23 months on the day of the first study visit ("12 to 23 months" means from the 12th month after birth to the day before the 24th month after birth).
* Informed consent form (ICF) had been signed and dated by the parent(s)/legally acceptable representative(s) and by an independent witness if required by local regulations.
* Participant and parent/legally acceptable representative were able to attend all scheduled visits and complied with all trial procedures.

Exclusion criteria:

* Participation in the 4 weeks (28 days) preceding the study vaccination or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the trial vaccination or planned receipt of any vaccine prior to Visit 2 except for influenza vaccination, which might be received at least 2 weeks before or after study vaccines. This exception included monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (i.e., mono- or polyvalent, polysaccharide, or Conjugate meningococcal vaccine containing serogroups A, C, W, or Y; or meningococcal B vaccine).
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically
* At high risk for meningococcal infection during the trial (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants travelling to countries with high endemic or epidemic disease).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances .
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine.
* Personal history of Guillain-Barré syndrome.
* Thrombocytopenia, as reported by the parent/ legally acceptable representative or suspected thrombocytopenia contraindicating intramuscular vaccination in the Investigator's opinion.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination in the Investigator's opinion.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature >= 38.0 degree Celsius). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 707 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (29):
- Denmark (3):
  - Investigational Site Number 2080001, Aarhus
  - Investigational Site Number 2080002, Hvidovre
  - Investigational Site Number 2080003, Odense
- Finland (9):
  - Investigational Site Number 2460006, Espoo
  - Investigational Site Number 2460005, Helsinki
  - Investigational Site Number 2460004, Jarvenpaa
  - Investigational Site Number 2460008, Kokkola
  - Investigational Site Number 2460007, Oulu
  - Investigational Site Number 2460003, Pori
  - Investigational Site Number 2460010, Seinäjoki
  - Investigational Site Number 2460001, Tampere
  - Investigational Site Number 2460002, Turku
- Germany (17):
  - Investigational Site Number 2760015, Bönnigheim
  - Investigational Site Number 2760004, Bramsche
  - Investigational Site Number 2760019, Bretten
  - Investigational Site Number 2760002, Erfurt
  - Investigational Site Number 2760017, Hamburg
  - Investigational Site Number 2760020, Herxheim
  - Investigational Site Number 2760007, Hürth
  - Investigational Site Number 2760013, Itzehoe
  - Investigational Site Number 2760011, Mannheim
  - Investigational Site Number 2760003, Mönchengladbach
  - Investigational Site Number 2760005, Mönchengladbach
  - Investigational Site Number 2760006, Schönau
  - Investigational Site Number 2760008, Schwaigern
  - Investigational Site Number 2760009, Schweigen
  - Investigational Site Number 2760018, Tauberbischofsheim
  - Investigational Site Number 2760010, Tuttlingen
  - Investigational Site Number 2760012, Wolfsburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: MEQ00065 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25309&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in 29 active centers in Denmark, Germany and Finland from 12 September 2019 to 03 September 2020.
Pre-assignment Details: A total of 707 participants were enrolled and randomized in the study.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Nimenrix® Vaccine | Group 3: NeisVac-C® Vaccine
Started | 232 | 235 | 240
Safety Analysis Set (All participants who had received one dose of study vaccine and analyzed according to the vaccine they actually received.) | 230 | 232 | 239
Completed | 228 | 229 | 239
Not Completed | 4 | 6 | 1
Not completed — Withdrawal by parent/guardian | 1 | 3 | 0
Not completed — Protocol deviation | 2 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Nimenrix® Vaccine | Group 3: NeisVac-C® Vaccine | Total
Number analyzed (Participants) | 232 | 235 | 240 | 707
Age, Continuous [Mean (Standard Deviation); unit: months] | 16.5 (3.27) | 16.6 (3.48) | 16.7 (3.45) | 16.6 (3.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 108 | 109 | 332
  Male | 117 | 127 | 131 | 375
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 225 | 226 | 236 | 687
  More than one race | 3 | 5 | 1 | 9
  Unknown or Not Reported | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Antibody Titers >=1:8 Against Meningococcal Serogroup C Measured by Serum Bactericidal Assay Using Human Complement (hSBA) Following Vaccination With MenACYW Conjugate Vaccine or Nimenrix® (Non-inferiority Analysis)
Description: Antibody titers against Meningococcal Serogroup C were measured by hSBA.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on hSBA per-protocol analysis set (PPAS) which was a subset that included all participants who received at least 1 dose of the study vaccine and had a valid post-vaccination serology result. The participants who presented protocol deviations were excluded from PPAS. Data for this outcome measure was planned to be collected and analyzed only for Group 1 and 2, and not for Group 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Nimenrix® Vaccine
Number analyzed (Participants) | 214 | 211
percentage of participants | 99.5 [97.4 to 100] | 89.1 [84.1 to 93.0]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Nimenrix® Vaccine; Test type: Non-Inferiority — The two-sided 97.5 percent (%) confidence interval (CI) was calculated based on the Wilson score method without continuity correction. The non-inferiority was demonstrated if the lower limit of the 97.5% CI of the percentage difference between compared groups was greater than (>) -10%; Difference in Percentage = 10.43, 97.5% CI 2-sided [5.68 to 16.2]

2. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Meningococcal Serogroup C Measured by hSBA Following Vaccination With MenACYW Conjugate Vaccine or Nimenrix® (Non-inferiority Analysis)
Description: GMT titers against Meningococcal Serogroup C were measured by hSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on hSBA PPAS which was a subset that included all participants who received at least 1 dose of the study vaccine and had a valid post-vaccination serology result. The participants who presented protocol deviations were excluded from PPAS. Data for this outcome measure was planned to be collected and analyzed only for Group 1 and 2, and not for Group 3.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Nimenrix® Vaccine
Number analyzed (Participants) | 214 | 211
titers | 515 [450 to 591] | 31.6 [26.5 to 37.6]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Nimenrix® Vaccine; Test type: Non-Inferiority — The two-sided 97.5% CI of the ratio of post-vaccination GMTs was calculated using normal approximation of log-transformed titers. The non-inferiority was demonstrated if the lower limit of the two-sided 97.5% CI of the ratio of GMTs between compared groups was >1/1.5; GMT Ratio = 16.3, 97.5% CI 2-sided [12.7 to 21.0]

3. Primary Outcome: GMTs of Antibodies Against Meningococcal Serogroup C Measured by hSBA Following Vaccination With MenACYW Conjugate Vaccine or Nimenrix® (Superiority Analysis)
Description: GMT titers against Meningococcal Serogroup C were measured by hSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 30 (post-vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Nimenrix® Vaccine
Number analyzed (Participants) | 214 | 211
titers | 515 [450 to 591] | 31.6 [26.5 to 37.6]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Nimenrix® Vaccine; Test type: Superiority — The two-sided 97.5% CI of the ratio of post-vaccination GMTs was calculated using normal approximation of log-transformed titers. The superiority was demonstrated if the lower limit of the two-sided 97.5% CI of the ratio of GMTs between compared groups was >1; GMT Ratio = 16.3, 97.5% CI 2-sided [12.7 to 21.0]

4. Primary Outcome: Percentage of Participants With Antibody Titers >=1:8 Against Meningococcal Serogroup C Measured by hSBA Following Vaccination With MenACYW Conjugate Vaccine or Nimenrix® (Superiority Analysis)
Description: Antibody titers against Meningococcal Serogroup C were measured by hSBA.
Time Frame: Day 30 (post-vaccination)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Nimenrix® Vaccine
Number analyzed (Participants) | 214 | 211
percentage of participants | 99.5 [97.4 to 100] | 89.1 [84.1 to 93.0]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Nimenrix® Vaccine; Test type: Superiority — The two-sided 97.5% CI was calculated based on the Wilson score method without continuity correction. The superiority was demonstrated if the lower limit of the 97.5% CI of the percentage difference between compared groups was >0%; Difference in Percentage = 10.43, 97.5% CI 2-sided [5.68 to 16.20]

5. Primary Outcome: Percentage of Participants With Antibody Titers >=1:8 Against Meningococcal Serogroup C Measured by Serum Bactericidal Assay Using Baby Rabbit Complement (rSBA) Following Vaccination With MenACYW Conjugate Vaccine or NeisVac-C® (Non-inferiority Analysis)
Description: Antibody titers against Meningococcal Serogroup C were measured by rSBA.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on rSBA PPAS which was a subset that included all participants who received at least 1 dose of the study vaccine and had a valid post-vaccination serology result. The participants who presented protocol deviations were excluded from PPAS. Data for this outcome measure was planned to be collected and analyzed only for Group 1 and 3, and not for Group 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 3: NeisVac-C® Vaccine
Number analyzed (Participants) | 213 | 215
percentage of participants | 100 [98.3 to 100] | 100 [98.3 to 100]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 3: NeisVac-C® Vaccine; Test type: Non-Inferiority — The two-sided 97.5% CI was calculated based on the Wilson score method without continuity correction. The non-inferiority was demonstrated if the lower limit of the 97.5% CI of the percentage difference between compared groups was >-10%; Difference in Percentage = 0.00, 97.5% CI 2-sided [-2.30 to 2.28]

6. Primary Outcome: GMTs of Antibodies Against Meningococcal Serogroup C Measured by rSBA Following Vaccination With MenACYW Conjugate Vaccine or NeisVac-C® (Non-inferiority Analysis)
Description: GMT titers against Meningococcal Serogroup C were measured by rSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 30 (post-vaccination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 3: NeisVac-C® Vaccine
Number analyzed (Participants) | 213 | 215
titers | 2143 [1870 to 2456] | 1624 [1425 to 1850]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 3: NeisVac-C® Vaccine; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMT Ratio = 1.32, 97.5% CI 2-sided [1.06 to 1.64]

7. Primary Outcome: GMTs of Antibodies Against Meningococcal Serogroup C Measured by rSBA Following Vaccination With MenACYW Conjugate Vaccine or NeisVac-C® (Superiority Analysis)
Description: GMT titers against Meningococcal Serogroup C were measured by rSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 30 (post-vaccination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 3: NeisVac-C® Vaccine
Number analyzed (Participants) | 213 | 215
titers | 2143 [1870 to 2456] | 1624 [1425 to 1850]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 3: NeisVac-C® Vaccine; Test type: Superiority — [test comment as in outcome 3, analysis 1]; GMT Ratio = 1.32, 97.5% CI 2-sided [1.06 to 1.64]

8. Secondary Outcome: Percentage of Participants With Antibody Titers >=1:8 Against Meningococcal Serogroup C Measured by rSBA Following Vaccination With MenACYW Conjugate Vaccine or Nimenrix® (Non-inferiority Analysis)
Description: Antibody titers against Meningococcal Serogroup C were measured by rSBA.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on rSBA PPAS which was a subset that included all participants who received at least 1 dose of the study vaccine and had a valid post-vaccination serology result. The participants who presented protocol deviations were excluded from PPAS. Data for this outcome measure was planned to be collected and analyzed only for Group 1 and 2, and not for Group 3.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Nimenrix® Vaccine
Number analyzed (Participants) | 213 | 210
percentage of participants | 100 [98.3 to 100] | 94.8 [90.8 to 97.4]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Nimenrix® Vaccine; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Difference in Percentage = 5.24, 97.5% CI 2-sided [1.83 to 9.85]

9. Secondary Outcome: GMTs of Antibodies Against Meningococcal Serogroup C Measured by rSBA Following Vaccination With MenACYW Conjugate Vaccine or Nimenrix® (Non-inferiority Analysis)
Description: GMT titers against Meningococcal Serogroup C were measured by rSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 30 (post-vaccination)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Nimenrix® Vaccine
Number analyzed (Participants) | 213 | 210
titers | 2143 [1870 to 2456] | 315 [252 to 395]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Nimenrix® Vaccine; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMT Ratio = 6.80, 97.5% CI 2-sided [5.04 to 9.18]

10. Secondary Outcome: GMTs of Antibodies Against Meningococcal Serogroup C Measured by rSBA Following Vaccination With MenACYW Conjugate Vaccine or Nimenrix® (Superiority Analysis)
Description: GMT titers against Meningococcal Serogroup C were measured by rSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 30 (post-vaccination)
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Nimenrix® Vaccine
Number analyzed (Participants) | 213 | 210
titers | 2143 [1870 to 2456] | 315 [252 to 395]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: Nimenrix® Vaccine; Test type: Superiority — [test comment as in outcome 3, analysis 1]; GMT Ratio = 6.80, 97.5% CI 2-sided [5.04 to 9.18]

11. Secondary Outcome: Percentage of Participants With Antibody Titers >=1:8 Against Meningococcal Serogroup C Measured by hSBA Following Vaccination With MenACYW Conjugate Vaccine or NeisVac-C® (Non-inferiority Analysis)
Description: Antibody titers against Meningococcal Serogroup C were measured by hSBA.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on hSBA PPAS which was a subset that included all participants who received at least 1 dose of the study vaccine and had a valid post-vaccination serology result. The participants who presented protocol deviations were excluded from PPAS. Data for this outcome measure was planned to be collected and analyzed only for Group 1 and 3, and not for Group 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 3: NeisVac-C® Vaccine
Number analyzed (Participants) | 214 | 216
percentage of participants | 99.5 [97.4 to 100] | 99.5 [97.4 to 100]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 3: NeisVac-C® Vaccine; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Difference in Percentage = -0.00, 97.5% CI 2-sided [-2.71 to 2.67]

12. Secondary Outcome: GMTs of Antibodies Against Meningococcal Serogroup C Measured by hSBA After Vaccination With MenACYW Conjugate Vaccine or NeisVac-C® (Non-inferiority Analysis)
Description: GMT titers against Meningococcal Serogroup C were measured by hSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 30 (post-vaccination)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 3: NeisVac-C® Vaccine
Number analyzed (Participants) | 214 | 216
titers | 515 [450 to 591] | 227 [198 to 260]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 3: NeisVac-C® Vaccine; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; GMT Ratio = 2.27, 97.5% CI 2-sided [1.82 to 2.84]

13. Secondary Outcome: GMTs of Antibodies Against Meningococcal Serogroup C Measured by hSBA Following Vaccination With MenACYW Conjugate Vaccine or NeisVac-C® (Superiority Analysis)
Description: GMT titers against Meningococcal Serogroup C were measured by hSBA. Titers were expressed in terms of 1/dilution.
Time Frame: Day 30 (post-vaccination)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 3: NeisVac-C® Vaccine
Number analyzed (Participants) | 214 | 216
titers | 515 [450 to 591] | 227 [198 to 260]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 3: NeisVac-C® Vaccine; Test type: Superiority — [test comment as in outcome 3, analysis 1]; GMT Ratio = 2.27, 97.5% CI 2-sided [1.82 to 2.84]

ADVERSE EVENTS:
Time Frame: Unsolicited adverse events (AEs) data were collected from Day 0 (pre-vaccination) up to Day 30 (post-vaccination). The solicited reactions were collected within 7 days post-vaccination. Serious AEs data were collected up to 30 days post-vaccination.
Description: Analysis was performed on Safety Analysis Set which included all participants who had received one dose of study vaccine and were analyzed according to the vaccine they actually received.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Nimenrix® Vaccine | Group 3: NeisVac-C® Vaccine
All-Cause Mortality (participants affected / at risk) | 0/230 | 0/232 | 0/239
Serious Adverse Events (participants affected / at risk) | 1/230 | 1/232 | 2/239
Other Adverse Events (participants affected / at risk) | 197/230 | 192/232 | 203/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=230) | Group 2: Nimenrix® Vaccine (N=232) | Group 3: NeisVac-C® Vaccine (N=239)
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Foreign Body In Throat (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=230) | Group 2: Nimenrix® Vaccine (N=232) | Group 3: NeisVac-C® Vaccine (N=239)
Diarrhoea (Gastrointestinal disorders) | 12 (14) | 14 (18) | 12 (12)
Teething (Gastrointestinal disorders) | 21 (22) | 11 (15) | 14 (19)
Toothache (Gastrointestinal disorders) | 16 (20) | 6 (6) | 7 (8)
Vomiting (Gastrointestinal disorders) | 20 (23) | 20 (20) | 16 (16)
Crying (General disorders) | 72 (73) | 73 (73) | 81 (82)
Injection Site Erythema (General disorders) | 85 (85) | 95 (95) | 95 (95)
Injection Site Pain (General disorders) | 96 (96) | 73 (73) | 91 (91)
Injection Site Swelling (General disorders) | 33 (33) | 34 (34) | 42 (42)
Pyrexia (General disorders) | 38 (41) | 43 (45) | 45 (47)
Nasopharyngitis (Infections and infestations) | 22 (22) | 19 (21) | 26 (26)
Rhinitis (Infections and infestations) | 10 (10) | 8 (8) | 14 (15)
Upper Respiratory Tract Infection (Infections and infestations) | 15 (15) | 11 (11) | 14 (14)
Decreased Appetite (Metabolism and nutrition disorders) | 59 (59) | 67 (67) | 67 (67)
Somnolence (Nervous system disorders) | 40 (40) | 41 (41) | 49 (49)
Irritability (Psychiatric disorders) | 101 (103) | 101 (101) | 107 (109)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 9 (10) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT03890367/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT03890367/SAP_001.pdf